CLINICAL TRIAL: NCT01094379
Title: A Randomised Comparison of Postoperative Pain and Recovery Between Single Incision Laparoscopic Cholecystectomy Using One Port and Standard Laparoscopic Cholecystectomy Using Four Ports
Brief Title: A Randomised Comparison Between Single Incision Laparoscopic Cholecystectomy and Standard Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Antonios Vezakis, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aretaieion01
Record Dates: First submitted 2010-03-23; First posted 2010-03-26 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: cholecystectomy; laparoscopic; pain; single incision
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard lap chole (Active Comparator): Laparoscopic cholecystectomy using four entry sites to the abdominal cavity
  Interventions: Procedure: Standard laparoscopic cholecystectomy
- Single incision lap chole (Active Comparator): Laparoscopic cholecystectomy using one entry site to the abdominal cavity
  Interventions: Procedure: Single incision laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Standard laparoscopic cholecystectomy — Laparoscopic cholecystectomy using four entry sites to the abdominal cavity
  Other Names: Traditional laparoscopic cholecystectomy
  Arms: Standard lap chole
Procedure: Single incision laparoscopic cholecystectomy — Laparoscopic cholecystectomy using one entry site to the abdominal cavity
  Other Names: One port laparoscopic cholecystectomy
  Arms: Single incision lap chole

SUMMARY:
Laparoscopic cholecystectomy has been established as the treatment of choice for symptomatic gallstone disease. The main advantages of laparoscopic surgery are the cosmetic result, reduced postoperative pain, shorter hospital stay and rapid return to normal activity. Although reduced, however, pain is still substantial and constitutes the main clinical problem after laparoscopic cholecystectomy, especially for planned day case procedures.

Recently, a new technique of laparoscopic cholecystectomy has been developed, in which all instruments are inserted through the same umbilical incision. The single incision laparoscopic surgery (SILS) technique for cholecystectomy has been proved to be feasible and safe by several studies.

The purpose of the study is to compare postoperative pain and operating time, nausea, vomiting, tissue damage, pulmonary function, cosmetic result, quality of life between SILS and standard laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy has been established as the treatment of choice for symptomatic gallstone disease. The main advantages of laparoscopic surgery are the cosmetic result, reduced postoperative pain, shorter hospital stay and rapid return to normal activity. Although reduced, however, pain is still substantial and constitutes the main clinical problem after laparoscopic cholecystectomy, especially for planned day case procedures.

Recently, a new technique of laparoscopic cholecystectomy has been developed, in which all instruments are inserted through the same umbilical incision. The single incision laparoscopic surgery (SILS) technique for cholecystectomy has been proved to be feasible and safe by several studies. However, there is not for the moment any randomized study between standard and SILS cholecystectomy published.

The primary end point of the study is to compare postoperative pain and secondary end points operating time, nausea, vomiting, tissue damage, pulmonary function, cosmetic result and quality of life.

Patients admitted for laparoscopic cholecystectomy to Aretaieion Hospital, under the care of four surgeons, will be entered into the study after signed consent is obtained. Randomization will be carried out preoperatively using blocks of random numbers. Anaesthesia will be standardized.

The same waterproof dressings, at the same sites, will be applied in all patients in order to prevent nursing and other staff from knowing what variant of operation has been carried out.

Postoperatively, all patients will receive and identical protocol of care. Postoperative pain will be assessed using a visual analogue pain score. The same analgesia will be prescribed in all the patients, if required. Postoperative analgesia, nausea or vomiting will be recorded.

Pulmonary function tests will be measured, in the sitting position, using a spirometer before and after the operation.

Tissue damage will be assessed by measuring CRP and Interleukin-6 (IL-6). Injury or inflammation of the human body results in increased concentrations of the acute-phase reactant proteins. CRP is very consistent in response and is, therefore, the most satisfactory single screening test for an acute phase reactant. IL-6 is one of the most important mediators of the acute phase response. It is secreted by T cells and macrophages to stimulate immune response to trauma.

The cosmetic result will be assessed by the patient.

Quality-of-life will be assessed using the EuroQoL EQ-5D questionnaire preoperatively and at 1 week postoperatively. The EQ-5D questionnaire is a generic measure of the quality of life, in which health status is defined in terms of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

Reevaluation of the patients will take place 1 week and 4 weeks after the operation in the outpatient clinic.

If we consider that we reduce postoperative pain at 35%, then with α: 0.05 and β: 0.20 we need 20 patients in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic cholelithiasis, admitted for laparoscopic cholecystectomy

Exclusion Criteria:

* Patients with acute cholecystitis
* Patients with extensive upper abdominal incisions
* Patients with body mass index >30
* Patients on regular analgesic medication

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24h
  Postoperative pain will be assessed using a visual analogue pain score

SECONDARY OUTCOMES:
operating time | Duration of surgical procedure
nausea or vomiting | 24 h
tissue damage | 24h
pulmonary function | 24h
cosmetic result | 4 weeks
Quality of life questionnaire | 1 week
  Quality-of-life will be assessed using the EuroQoL EQ-5D questionnaire preoperatively and 1 week postoperatively. The EQ-5D questionnaire is a generic measure of the quality of life, in which health status is defined in terms of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Vezakis, lecturer, Principal Investigator — University of Athens
Locations (1):
- Academic Department of Surgery, Aretaieion Hospital, Athens, Greece

REFERENCES:
- [Background] Tacchino R, Greco F, Matera D. Single-incision laparoscopic cholecystectomy: surgery without a visible scar. Surg Endosc. 2009 Apr;23(4):896-9. doi: 10.1007/s00464-008-0147-y. Epub 2008 Sep 25. PMID 18815836
- [Background] Chow A, Purkayastha S, Aziz O, Paraskeva P. Single-incision laparoscopic surgery for cholecystectomy: an evolving technique. Surg Endosc. 2010 Mar;24(3):709-14. doi: 10.1007/s00464-009-0655-4. Epub 2009 Aug 18. PMID 19688389
- [Derived] Steinemann DC, Raptis DA, Lurje G, Oberkofler CE, Wyss R, Zehnder A, Lesurtel M, Vonlanthen R, Clavien PA, Breitenstein S. Cosmesis and body image after single-port laparoscopic or conventional laparoscopic cholecystectomy: a multicenter double blinded randomised controlled trial (SPOCC-trial). BMC Surg. 2011 Sep 12;11:24. doi: 10.1186/1471-2482-11-24. PMID 21910897